CLINICAL TRIAL: NCT04923971
Title: Safety and Performance Monitoring During Occupational Work II
Acronym: COBRAII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Biotechnology High Performance Computing Software Applications Institute (Unknown)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H21-0016
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Intervention Model Description: Participants will perform hand-dexterity tasks in three different ambient temperatures 1) 0C 2) -10C, and 3) -20C surrogate (-10C with 3m/s wind speed to simulate -20C conditions)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0C Trial (Active Comparator): Participants will be sitting in a chair performing hand dexterity tasks in 0C (32F) conditions. Total rest period is 2 hours. After 2 hours, participants will perform athletic performance related tasks consisting of agility, power, muscular strength, and aerobic fitness.
  Interventions: Other: Purdue Pegboard
- -10C Trial (Active Comparator): Participants will be sitting in a chair performing hand dexterity tasks in -10C (14F) conditions.Total rest period is 2 hours. After 2 hours, participants will perform athletic performance related tasks consisting of agility, power, muscular strength, and aerobic fitness.
  Interventions: Other: Purdue Pegboard
- -20C Surrogate Trial (Active Comparator): Participants will be sitting in a chair performing hand dexterity tasks in -10C + 3m/s wind (14F+6 mph wind) conditions. Total rest period is 2 hours. After 2 hours, participants will perform athletic performance related tasks consisting of agility, power, muscular strength, and aerobic fitness.
  Interventions: Other: Purdue Pegboard

INTERVENTIONS:
Other: Purdue Pegboard — Participants will assemble the pegboard with their left, right, and both hands in each environmental condition.

SUMMARY:
BHSAI is developing a computational system that provides early alerts of a rise and fall in core body temperature to help reduce the risk of thermal injury in the field and during training. The goal of the body temperature alerting system is to use it during rest, exercise in the heat and cold. Therefore, the primary purpose of this investigation is to validate a body temperature alerting system using physiological responses that occur during rest and exercise in different cold environments. Multiple cold ambient temperatures will be validated.

DETAILED DESCRIPTION:
This study will employ a randomized, cross-over design to assess the effect of three different cold ambient temperatures on skin temperature at peripheral regions, core temperature (rectal), metabolic heat production, hand dexterity measures at rest, and athletic performance assessment after rest in cold ambient temperatures. The three different trials for this study will include ambient temperatures at: A. 0°C (32°F), B. -10°C (14°F), and C. Surrogate -20°C (-10°C + 3 m/s wind speed [14°F + 6 mph]). This will be accomplished by use of a environmental chamber.

Participants will be assigned after medical clearance is granted. Visit specific information is described below, however, specific data collection protocols for dependent variables and procedures are included below the description of the study design. Participants will be asked to sign a photo/video release form to be used in research projects, scientific publications/conferences and for educational purposes. Participants may be videoed or photographed while exercising or resting in the environmental chamber.

During the 0°C (32°F) and -10°C (14°F) trials, participants will wear cold weather gear as described by BHSAI. All cold weather gear will be machine-washable, provided to the participants and properly fitted to each individual. Clothing will be kept in the laboratory, machine-washed by manufacturer recommendations. Participants will not be able to keep clothing used upon completion of the study. These trials will also have a wind speed of 1 m/s. For the surrogate -20°C (-4°F) experiment, ambient temperature will be -10°C (14°F) with wind speed approximately at 3 m/s (6 mph) to serve as an aggregate for -20°C (-4°F). Wind will not be facing the participant. Participants will wear all cold weather gear listed above with the exception of the microfleece cap and shell layer for hand (Figure 2). For all trials, participants will rest upright on a chair with feet above the ground and hands on the arms of the chair (exposed to air). The participant will remain seated for 120 minutes. For additional safety of the participants, the experiment will be terminated if the core body temperature falls below 35°C (95°F) and/or the skin temperature in any of the peripheral regions falls below 8°C (46°F). During the three testing sessions, the participants will wear a Samsung Gear S3 smartwatch on their non-dominant arm and a Polar chest strap. These devices would be paired with a Samsung Galaxy Note 4 smartphone that runs the 2B-Cool algorithm for core temperature estimation using data from the smartwatch. These devices will be used in conjunction with data from the rectal and skin temperature sensors to validate the sponsors' temperature prediction algorithm. All devices will be cleaned prior to and after participant use per manufacturer instructions. These devices would be provided by BHSAI to the University of Connecticut. During the three testing sessions, in addition to the BHSAI-provided devices, participants will wear thermistors to record the skin temperature (finger-tip and base of finger, hand dorsum, big toe, nose, cheek, ear tip, chin, and forehead and will privately insert a rectal thermometer 15 cm (~4-6 ins) beyond the anal sphincter to record the gold-standard core temperature.VO2 data will also be assessed to collect metabolic heat production. Hand dexterity will be assessed using the validated Purdue pegboard test.

During all three sessions, researchers will ensure that the smartwatch is placed approximately 1-inch proximal to the wrist and fits snuggly to ensure accurate heart-rate measurements. Researchers will also ensure that the devices are paired with the smartphone and the physiological variables are being recorded on the phone before commencement of the session. Since different devices will be used for measuring the physiological variables and the associated gold standard, researchers will record the starting time-stamp from the smartphone and the gold-standard recording computer to ensure time synchronization.

Following the 120-minute seated rest period, a performance battery will be utilized to assess athletic performance in 3 different cold environments. Agility/reaction time, power, muscular strength, sprint performance on a cycle ergometer, and 1-mile time trial on a motorized treadmill will be assessed. An environmental symptom questionnaire (ESQ) will be administered at the end of the performance battery prior to exiting the chamber. All trials will be approximately 3-4 hours each. Total participation in the study is approximately 12-14 hours of time for the participant.

Baseline Testing (Visit 1)

Participants who are approved to participate will be scheduled for baseline anthropometrics and VO2max testing visit. Prior to arrival to the lab, participants will be given instructions (Appendix K) on proper hydration practices, avoidance of alcohol and caffeine (24 and 12 hours, respectively). Participants will be allowed to consume their normal diet during the study. Participants will be required to take the Korey Stringer Institute COVID-19 Pre-Screening Questionnaire (Appendix J) remotely through Qualtrics. Upon arrival to the lab, participants will provide a urine sample in a clean urine cup. Key study personnel will determine participants urine color using a validated urine color chart by Armstrong et al.3 Urine specific gravity (USG) will also be assessed. Euhydration will be defined USG ≤1.020. Urine specific gravity and urine color will be assessed. Participants will only be permitted to continue to the VO2max test if the euhydrated criteria of a USG ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the participant will be asked to drink 500mL of water to ensure proper hydration status. Nude body mass will also be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room (Defender R7000 Xtreme; OHAUS Corp., Parsippany, NJ, USA). Weight will be recorded in kilograms. Participants will fill out a Karolinska Sleep Diary (Appendix I) prior to collecting anthropometrics. Height will be measured with a tape measure. Percent body fat will be measured using Air displacement plethysmography (BodPod®; Cosmed, Software Version 4.2+, Concord, CA, USA). This will take less than ~5 minutes to complete. Participants will also be asked to complete a maximal oxygen uptake (VO2max) test on a treadmill in a thermoneutral environment. This test will provide aerobic fitness levels of the participants. A heart rate monitor and strap will be given to the participants to wear during the VO2max test. A metabolic mask will be used in order to determine RER. When the participant is ready, the test will begin. This test begins at a speed equivalent to a jog at 2% grade and the speed incrementally rises every 2 minutes until the participant reaches volitional fatigue. Maximal oxygen consumption, respiratory exchange ratio (RER), heart rate, and rating of perceived exertion (RPE) will be collected throughout this test. This test will take approximately 20 minutes. After VO2max testing, researchers will familiarize the participant with the hand dexterity test and the performance battery. Agility/reaction time, power, muscular strength, sprint performance on a cycle ergometer, and 1-mile time trial. Additionally, participants will be familiarized with all scales (RPE, thermal sensation scale, thirst scale, fatigue scale, and environmental symptom questionnaire [ESQ]) during this session (Appendix C). Scheduling will be completed for each participant prior to discharge from the Baseline familiarization visit. This visit will take approximately 1-2 hours.

Trial Day Procedures (All 3 Cold Temperature Trials)

Participants will be allowed to make-up trial visits if they are sick, suffer an injury or do not meet hydration requirements. Participants will be asked if they have a current illness or taking medications to determine whether they can complete the trial. The participant's visit will be rescheduled if they have a fever, current illness or taking medications that influence body temperature. If the participant indicates they have had a COVID-19 exposure prior to any scheduled trial, they will be required to follow University protocols and acquire a negative test result in order to remain eligible for the study. Trials will be on separate days at least 3 days apart.

Participants will be allowed to consume their normal diets prior to all visits. Upon arrival to the lab, participants will also be asked to indicate if they have consumed alcohol or caffeine in the last 24 hours and 12 hours, respectively. They will not be asked to specify exactly what they have consumed, but if they provide a positive indication, their trial will be rescheduled for another day. The participants will also be asked to complete a subjective sleep questionnaire as the arrive to the lab. Next, participants will provide a urine sample in a clean urine cup. Urine specific gravity and urine color will be assessed. Nude body mass will be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Hydration status of each participant will also be addressed prior to entering and exiting the chamber. Participants will only be permitted to continue to the trial if the euhydrated criteria of a urine specific gravity (USG) ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the participant will be asked to drink 500 mL of water to ensure proper hydration status. Participants will be given instructions at the prior visit about how to obtain desired hydration status for the upcoming trial.

Participants will privately insert a rectal thermometer 15 cm beyond the anal sphincter and wear a heart rate monitor strap. Additionally, participants will wear 9-site skin temperature sensors (Biopac, see diagram below skin temperature). Key personnel will apply the skin temperature sensors with medical tape to the participants' finger-tip and base of finger, hand dorsum, big toe, nose, cheek, ear tip, chin, and forehead. Participants will also have 4 iButton skin temperature sensors placed on four locations (shoulder, chest, calf, thigh) to assess mean skin temperature. The participants will wear a Samsung Gear S3 smartwatch on their non-dominant arm and a heart-rate monitor chest strap. These devices would be paired with a Samsung Galaxy Note 4 smartphone that runs the 2B-Cool algorithm for core temperature estimation using data from the smartwatch. These devices will be provided by BHSAI to the University of Connecticut. Participants will then don the cold-environment clothing (purchased from grant funding), described previously, before entering the chamber. VO2 data will also be assessed to collect metabolic heat production. Participants will rest in a lounge chair for 2 hours with hand-dexterity tests performed every 30 minutes. All participants will drink ad libitum throughout all trials.. Following the 120-minute seated rest period, a performance battery will be utilized to assess athletic performance in 3 different cold environments: Agility/reaction time, power, muscular strength, sprint performance on a cycle ergometer and 1-mile time trial. USG and urine color and will be assessed prior to the discharge of the participant from the laboratory. These visits will take approximately 3-4 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Males between the ages of 18-28 years
2. Have been cleared to participate by the medical monitor for this study
3. Must perform aerobic exercise for 150 minutes per week.

Exclusion Criteria:

1. Are a female
2. Have a history of adverse reaction to the cold environments, such as cold urticaria (i.e.

   allergy to the cold) and/or Raynaud's phenomenon [disorder that causes decreased blood flow to peripheral body parts (e.g. fingers and toes)]
3. Identify any symptoms of COVID-19, which include:

   1. Fever that exceeds 100.4F
   2. New loss of smell and/or taste
   3. Cough
   4. Shortness of breath/difficulty breathing
   5. Chills
   6. Muscle pain
   7. Fatigue
   8. Headache
   9. Sore throat
4. Tested positive for COVID-19 within the past 6 months.
5. Have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.
6. Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally).
7. Other current illnesses at time of testing
8. History of cardiovascular, metabolic, chronic respiratory disease, peripheral arterial disease, or coagulopathy.
9. Currently taking a medication that is known to influence body temperature or blood flow (amphetamines, antihypertensives, anticholinergics, acetaminophen, diuretics, NSAIDs, aspirin, vasoactive medications)
10. Currently smoking (cigarettes, vaporizers, e-cigarettes)
11. Have a history of claustrophobia
12. Have a history of allergic reactions to medical tape
13. Hypothyroidism
14. History of or current eating disorder(s)
15. Are anemic

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender women, Transgender men, and transgender women are excluded from the current study because the sponsor of the study has requested that this testing be done in physically active cisgender males. It is assumed that they either currently have data on women or transgender women/men to compare this to or have a strategic initiative from a marketing or business perspective that only involves cisgender men.
Enrollment: 15 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Rectal Temperature | Measured continuously during one, 120 min rest blocks and 1 20-30 min athletic performance test period.]
  Rectal thermometer will be self-inserted by participant to assess core temperature
Change in Heart Rate | Measured continuously during one, 120 min rest block and 1 20-30 min athletic performance test period.]
  A heart rate monitor will be worn by participant throughout the rest period and performance battery protocol
Change in Mean Skin temperature | Measured continuously during one, 120 min rest block and 1 20-30 min athletic performance test period.]
  Prior to the start of the protocol, participants will be instrumented with 9-site (Biopac) and 4-site mean skin temperature (iButton) sensors. The Biopac skin temperature sensors will be placed on the finger-tip and base of finger, hand dorsum, big toe, nose, cheek, ear tip, chin, and forehead. The iButton skin temperature sensors will be placed on the chest, arm, thigh, and calf.

SECONDARY OUTCOMES:
Change in Rating of Perceived Exertion | Measured during 1 20-30 min athletic performance test period
  The Rating of Perceived Exertion (RPE) uses a Borg Scale (scored 6-20) that indicates how hard the participant feels they are working. 6 represents rest and 20 represents maximal exertion. A high score indicates more perceived exertion.
Change in Thermal Sensation | Every 5 minutes of the rest block (120 mins) and 1 athletic performance battery (20-30 mins)
  0-8 Scale (cold to hot) that indicated how cold or hot the participate feels. 0 = extremely cold, 8 = extremely hot.
Change in Perception of Fatigue | Every 5 minutes of the rest block (120 mins) and 1 athletic performance battery (20-30 mins)
  0-10 (no fatigue to extreme fatigue) Scale that indicates how fatigued the participate feels. High score indicates more fatigue (negative outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Casa, Principal Investigator — Korey Stringer Institute, University of Connecticut
Locations (1):
- Korey Stringer Institute, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No